CLINICAL TRIAL: NCT01333085
Title: Phase I/II Study of Induction Chemotherapy With Weekly RAD001, Carboplatin and Paclitaxel in Unresectable or Inoperable Locally Advanced Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: Everolimus, Carboplatin, and Paclitaxel in Locally Advanced Head and Neck Cancer That Cannot Be Removed by Surgery
Acronym: CAPRA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000698330; FRE-GERCOR-CAPRA; FRE-GERCOR-O08-1; EU-21109; EUDRACT-2008-005702-39
Record Dates: First submitted 2011-04-08; First posted 2011-04-11 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2013-03

CONDITIONS: Head and Neck Cancer
Keywords: stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV verrucous carcinoma of the oral cavity; stage IV squamous cell carcinoma of the oropharynx; tongue cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms | interventions — Carboplatin; Everolimus; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RAD001-paclitaxel-carboplatin (Experimental): RAD001: 20,30 or 50 mg PO 9 weekly cycles Paclitaxel: 60 mg/m²IV, in 1 hour, 9 weekly cycles Carboplatin AUC2 IV in 1 hour,9 weekly cycles
  Interventions: Drug: carboplatin; Drug: RAD001; Drug: paclitaxel

INTERVENTIONS:
Drug: carboplatin
Drug: RAD001
  Other Names: everolimus
Drug: paclitaxel

SUMMARY:
RATIONALE: Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase I/II trial is studying the side effects and best dose of giving everolimus together with carboplatin and paclitaxel in treating patients with locally advanced head and neck cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum-tolerated dose of everolimus when combined with carboplatin and paclitaxel in chemonaïve patients with unresectable or inoperable locally advanced head and neck squamous cell carcinoma. (Phase I)
* To determine the safety profile of weekly everolimus in combination with carboplatin and paclitaxel in chemonaïve patients with unresectable or inoperable locally advanced head and neck squamous cell carcinoma. (Phase I)
* To determine the anti-tumor activity of this regimen, in terms of objective response rate of the combination, according to the RECIST criteria in these patients. (Phase II)

Secondary

* To identify molecular markers of resistance to this regimen in these patients.
* To assess objective response rate before and after completion of radiation therapy in these patients. (Phase II)

OUTLINE: This is a multicenter, phase I dose-escalation study of everolimus followed by a phase II study.

* Phase I: Patients receive paclitaxel IV over 1 hour, carboplatin IV over 1 hour, and escalating doses of oral everolimus on days 1, 8, and 15. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity.
* Phase II: Patients receive paclitaxel and carboplatin as in phase I and oral everolimus (at a dose determined in the phase I portion of the study) on days 1, 8, and 15. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity.

After the completion of combination therapy, patients may receive radiotherapy or surgery, at the investigator's discretion.

Blood samples are collected for translational research and molecular markers analysis at baseline and weeks 1, 4, and 9. Tissue samples are collected at baseline and periodically during the study for biomarker and other laboratory analysis.

After completion of study treatment, patients are followed up at 14 days and periodically thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma of the oral cavity, oropharynx, larynx, or hypopharynx

  * Locally advanced disease (T4 N0-N3 disease)
  * Unresectable disease OR resectable disease with surgery contra-indication
  * No stage I, II, III, or IVc disease
* Measurable lesions defined as those accurately measured in ≥ 1 dimension (longest diameter to be recorded) as ≥ 20 mm with conventional techniques or as ≥ 10 mm with spiral CT scan
* No known brain metastases (cerebral CT scan is not required if no symptom is present)

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Life expectancy > 3 months
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL
* Total bilirubin ≤ 1.25 times upper limit of normal (ULN)
* Transaminases ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 5 times ULN
* Creatinine clearance ≥ 60 mL/min
* Glycemia ≤ 1.5 times ULN
* Cholesterol level ≤ 7.30 mmol/L
* Serum total protein normal
* Oxygen saturation > 88%
* Able to swallow pills
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* No preexisting neuropathy ≥ grade 2
* No uncontrolled disease including any of the following:

  * Diabetes
  * Hypertension
  * Symptomatic congestive heart or pulmonary failure
  * Renal or hepatic chronic disease
  * Severe infectious disease
* No active hemorrhagic syndrome
* No prior history of cancer within the past 5 years, except in situ cervical cancer and basal cell skin carcinoma
* No psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Registration in a national health care system (CMU included)
* Not eligible for organ preservation program

PRIOR CONCURRENT THERAPY:

* No prior therapy for this cancer
* No prior chemotherapy unless received for treatment of another primary tumor considered in remission
* No prior investigational drug
* More than 30 days since prior participation in another therapeutic trial
* No prior or concurrent radiotherapy (except anterior radiotherapy) unless received for treatment of another primary tumor considered in remission
* No concurrent CYP3A4 strong inhibitors (e.g., azole antimycotics [itraconazole, ketoconazole], HIV protease inhibitor [ritonavir], erythromycin, anti-epileptic drugs [phenytoin, carbamazepine])
* No concurrent anti-coagulant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2009-10; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | weekly
  to determine the maximum tolerated dose (MTD) and recommended dose of weekly RAD001 in combination with carboplatin and paclitaxel (phase I)
objective response rate | 9 weeks
  To access the objective response rate of the combination RAD001-carboplatin-Paclitaxel according the the RECIST criteria, after 9 weekly cycles (phase II)

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine Faivre, Principal Investigator — Hopital Beaujon
Locations (5):
- France (5):
  - Hopital Beaujon, Clichy
  - Centre Léon Berard, Lyon
  - Institut Curie, Paris
  - Hôpital Privé Saint Joseph, Paris
  - Institut Claudius Regaud, Toulouse